CLINICAL TRIAL: NCT05813860
Title: Preemptive HLADQA1*05 Genotyping for the Use of Infliximab in Chinese Crohn's Disease：A Multicenter, Prospective, Controlled, Randomized Study
Brief Title: HLADQA1*05 Genotype and the Efficacy of Treatment With Infliximab in Chinese Population Crohn's Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023ZSLYEC-123
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Crohn Disease; Infliximab
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Infliximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Infliximab monotherapy, the first dose of 5 mg/kg of this product is provided, followed by the same dose at weeks 2 and 6 after the first dose and every 8 weeks thereafter.
  Interventions: Drug: Infliximab
- Infliximab+azathioprine (Active Comparator): Infliximab was given in combination with azathioprine, and Infliximab dosing was the same as in the experimental group, with azathioprine at 1-2 mg/kg/d.
  Interventions: Drug: Azathioprine; Drug: Infliximab

INTERVENTIONS:
Drug: Azathioprine — azathioprine in combination with Infliximab, with a dose of 1-2 mg/kg/d.
  Arms: Infliximab+azathioprine
Drug: Infliximab — 5mg/kg for the first dose, and the same dose at weeks 2 and 6 after the first dose and every 8 weeks thereafter. Treatment with single Infliximab or combined azathioprine, respectively.

SUMMARY:
Crohn's disease (CD) is a chronic non-specific inflammatory disease of the intestine. Infliximab (IFX) is a kind of one of the anti-tumor necrosis factor agents (anti-TNF) and is the main clinical treatment drug for Crohn's disease, but approximately 30-50% of patients develop a secondary non-response to respond within one year. The main cause of secondary non-response failure is the formation of anti-IFX anti-drug antibodies (ADA). The human leukocyte antigen (HLA) gene is a complex allele that has been associated with susceptibility to a variety of diseases. Studies have shown that HLADQA1*05 allele carriage significantly increases the immunogenicity of anti-tumor necrosis factor agents (anti-TNF) and the risk of ADA formation, resulting in a significant reduction in the efficacy of IFX. Our previous retrospective study found an increased risk of ADA, IFX failure to respond and discontinuation in patients with HLADQA1*05 variants, and that IFX in combination with immunosuppression improved clinical outcomes in wild-type genotype patients, whereas combination therapy in patients with variant genotype did not optimize clinical outcomes significantly. Therefore, we believe that the impact of HLADQA1*05 on the efficacy of IFX in the Chinese population is unclear, and the combination of immunosuppressants in patients with variant HLADQA1*05 genotype remains to be validated due to insufficient sample size. We hypothesized that HLADQA1*05 wild-type CD patients would have better clinical remission when treated with IFX than HLADQA1*05 variant patients and that the combination of immunosuppressants would improve the outcome in wild-type patients but not in variant patients. By advancing this project, we hope to provide high quality evidence on the clinical use of IFX in Crohn's disease in the Chinese population and help physicians to be more selective in the use of IFX alone or in combination with azathioprine, or to switch treatment in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Crohn's disease who meet the diagnostic criteria of the Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Disease (Beijing, 2018)
* Meet the indications for IFX use
* CDAI score of 220-450; age≥18 years, regardless of gender
* Participants or family members able to understand the study protocol and willing to participate in this study by providing written informed consent

Exclusion Criteria:

* NUDT 15 CT and TT genotypes; previous treatment with IFX and/or other anti-TNF biologics
* Participants who are proposed to have given birth and/or breastfeeding in the 12 months
* those with immunosuppressive intolerance or contraindications
* concurrent chronic diseases or factors of other systems (including severe cardiopulmonary, hepatic and renal, neurological, psychiatric, rheumatic and immune diseases, alcoholism, drug dependence, other chronic active diseases and long-term hormonal or immunosuppressive drugs)
* Excluding infectious diseases (tuberculosis, etc.)
* Excluding tumor-related diseases (lymphoma, gastrointestinal tract tumors, etc.)
* any medical condition/combined surgery/medication/other clinically significant abnormal laboratory tests which, in the judgment of the investigator, may affect the results of the test
* Known refusal or inability to follow protocol requirements for any reason (including planned clinical visits and examinations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission without corticosteroid use at 102 weeks | 102 weeks
  CDAI score below 150 and no systemic corticosteroids at any dose or Budesonide ≥ 3 weeks.

SECONDARY OUTCOMES:
Clinical response at 14 weeks | 14 weeks
  Decrease in CDAI score ≥70 or CDAI score <150
Positive for ADA | 102 weeks
  Transient or persistent serum ADA concentration ≥ 10 AU/mL
IFX Intensive Therapy | 102 weeks
  Includes increased doses and shorter cycles due to the recurrence of disease
IFX Failure to Respond | 102 weeks
  Recurrence of disease during treatment with IFX with increased in CDAI score ≥ 70 or CDAI score ≥150
Adverse drug events | 102 weeks
  Allergies, infusion reactions, infections, tumors, liver damage, bone marrow suppression, hair loss, etc.
IFX discontinuation | 102 weeks
  Includes discontinuation due to IFX non-response or adverse events